CLINICAL TRIAL: NCT02143492
Title: Tumor Collection From Routine Nephrectomy for Subjects With Advanced Stage RCC
Status: Completed | Type: Observational
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: AGS-NTS-020
Record Dates: First submitted 2014-04-30; First posted 2014-05-21 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma; Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Excess kidney cancer tumor specimen
Oversight: Data Monitoring Committee: No

SUMMARY:
Standard treatment for kidney cancer is to remove the tumors from the body with surgery. The purpose of this clinical trial is to collect, preserve, and store excess kidney cancer tumor specimens that would normally be discarded after surgery.

DETAILED DESCRIPTION:
The purpose of this non-treatment, non-interventional protocol is to collect, preserve, and store excess tumor specimens, which would otherwise be discarded, following routine nephrectomy for subjects with advanced renal cell carcinoma (RCC). The collected tumor specimen will be preserved under current Good Manufacturing Practice conditions and will not be used for any other research or therapeutic purpose without a separate consent from the subject, specific to the intended use on a separate Institutional Review Board or Institutional Ethics Committee approved Argos sponsored study.

Following routine nephrectomy (partial or cytoreductive) as indicated for subjects with advanced RCC, small samples of the excised tumor will be sectioned and placed into an RNA preservative solution as supplied by the sponsor. After collection, this preserved tumor specimen will be shipped to a repository operating under current Good Manufacturing Practice conditions. The tumor specimen will be stored for no longer than five years unless subsequent consent is obtained for extended storage or other use.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years
* 2. Diagnosis or clinical signs of advanced RCC (Stage III or IV RCC; Refer to Appendix A)
* 3. Scheduled for cytoreductive or partial (unilateral or bilateral) nephrectomy
* 4. Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of tumor specimen collection prior to enrollment

Exclusion Criteria:

* 1. Evidence of brain metastases prior to nephrectomy
* 2. Requirement for systemic chronic immunosuppressive drugs or systemic chronic corticosteroids, for active autoimmune disorder(s) or other conditions (e.g.: rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, organ transplant recipient, etc.)
* 3. History of HIV infection, or history of chronic infection with Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with advanced renal cell carcinoma (kidney cancer)
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Tumor Specimen | 5 years
  Tumor specimen collection

CONTACTS AND LOCATIONS:
Overall Officials: Neal Shore, MD, FACP, Principal Investigator — Carolina Urologic Research Center
Locations (5):
- United States (5):
  - Englewood, Colorado
  - Marietta, Georgia
  - Woodbury, Minnesota
  - Rock Hill, North Carolina
  - Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No